CLINICAL TRIAL: NCT00745823
Title: A Phase III Multicenter, Double-Blind, Randomized, Active Comparator-Controlled Clinical Trial to Study the Safety and Efficacy of Once Daily Raltegravir (MK0518) Versus Twice Daily Raltegravir, Each in Combination With TRUVADA™, in Treatment-Naïve HIV Infected Patients
Brief Title: A Study to Determine the Safety and Efficacy of Once Daily Raltegravir Compared to Twice Daily Raltegravir (MK-0518-071)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Primary efficacy analysis at Week 48 did not demonstrate non-inferiority of raltegravir 800 mg once daily versus raltegravir 400 mg twice daily
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0518-071; 2008_543 (Other: Merck Registration Number); CTRI/2009/091/000145 (Registry Identifier: CTRI)
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Results first posted 2012-04-25 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-02

CONDITIONS: HIV
Keywords: HIV Infections; Treatment Naïve
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Raltegravir 400 mg b.i.d. (Active Comparator)
  Interventions: Drug: Comparator: Raltegravir 400 mg b.i.d.; Drug: TRUVADA™
- Raltegravir 800 mg q.d. (Experimental)
  Interventions: Drug: Experimental: Raltegravir 800 mg q.d.; Drug: TRUVADA™

INTERVENTIONS:
Drug: Comparator: Raltegravir 400 mg b.i.d. — Raltegravir 400 mg tablet by mouth (PO) twice daily (b.i.d.) + two raltegravir placebo tablets + one tablet of TRUVADA™ once daily (q.d.)
  Other Names: ISENTRESS™
  Arms: Raltegravir 400 mg b.i.d.
Drug: Experimental: Raltegravir 800 mg q.d. — Raltegravir 800 mg tablet PO q.d. + two raltegravir placebo tablets + one tablet TRUVADA™ q.d.
  Other Names: ISENTRESS™
  Arms: Raltegravir 800 mg q.d.
Drug: TRUVADA™ — One tablet TRUVADA™ q.d. (fixed combination 200 mg emtricitabine and 300 mg tenofovir disoproxil fumarate)

SUMMARY:
A study to evaluate the safety, tolerability and efficacy of once daily Raltegravir compared to twice daily raltegravir when each is given in combination with TRUVADA™ in treatment-naïve human immunodeficiency virus (HIV)-infected patients.

DETAILED DESCRIPTION:
Following the 96-week double-blind study period (MK0518-071)(NCT00745823), subjects may enroll in an extension study (MK0518-071-10)(NCT00745823). From weeks 96 to 120, subjects' treatment assignments will remain as in the base study.

From week 120 to 240, all subjects will receive open-label raltegravir (800 mg, once daily) in combination with TRUVADA™.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female 18 years of age or older
* Patient is HIV positive
* Patient is naïve to antiretroviral therapy (ART) or has received less than 7 days total of any ART

Extension Study:

* The planned extension study did not take place as the study was terminated after the Week 48 analysis.

Exclusion Criteria:

* Patient is a user of recreational or illicit drugs or has had a recent history (within the last year) of drug or alcohol abuse or dependence
* Patient has documented resistance to tenofovir or emtricitabine
* Patient is currently participating or has participated in a study with an investigational compound or device within 45 days of signing informed consent
* Patient is pregnant or breastfeeding, or expecting to conceive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 775 (Actual)
Dates: Start 2008-09; Primary Completion 2010-10 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Eron JJ Jr, Rockstroh JK, Reynes J, Andrade-Villanueva J, Ramalho-Madruga JV, Bekker LG, Young B, Katlama C, Gatell-Artigas JM, Arribas JR, Nelson M, Campbell H, Zhao J, Rodgers AJ, Rizk ML, Wenning L, Miller MD, Hazuda D, DiNubile MJ, Leavitt R, Isaacs R, Robertson MN, Sklar P, Nguyen BY; QDMRK Investigators. Raltegravir once daily or twice daily in previously untreated patients with HIV-1: a randomised, active-controlled, phase 3 non-inferiority trial. Lancet Infect Dis. 2011 Dec;11(12):907-15. doi: 10.1016/S1473-3099(11)70196-7. Epub 2011 Sep 18. PMID 21933752

RESULTS

PARTICIPANT FLOW:
Groups:
- Raltegravir 800 mg q.d.: Raltegravir 800 mg by mouth (PO) once daily (q.d.) plus placebo to raltegravir PO twice daily (b.i.d.) plus one tablet of TRUVADA™ for 96 weeks
- Raltegravir 400 mg b.i.d.: Raltegravir 400 mg PO b.i.d. plus placebo to raltegravir PO q.d. plus one tablet of TRUVADA™ for 96 weeks
Period: Overall Study
Arm/Group | Raltegravir 800 mg q.d. | Raltegravir 400 mg b.i.d.
Started | 386 | 389
TREATED Week 0 - 96 | 382 | 388
Completed | 1 | 3
Not Completed | 385 | 386
Not completed — Adverse Event | 5 | 3
Not completed — Lack of Efficacy | 20 | 6
Not completed — Lost to Follow-up | 10 | 11
Not completed — Physician Decision | 10 | 5
Not completed — Pregnancy | 0 | 4
Not completed — Withdrawal by Subject | 14 | 8
Not completed — Study Terminated by Sponsor | 326 | 349

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Raltegravir 800 mg q.d. | Raltegravir 400 mg b.i.d. | Total
Number analyzed (Participants) | 386 | 389 | 775
Age, Customized [Number; unit: participants]
  Between 18 and 64 years | 382 | 382 | 764
  >=64 years | 4 | 7 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 90 | 158
  Male | 318 | 299 | 617

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With HIV Ribonucleic Acid (RNA) <50 Copies/mL at 48 Weeks
Time Frame: Week 48
Population: Data were analyzed for all participants treated with study drug. Participants who did not complete the study were treated as treatment failures.
Measure: Number; unit: Participants
Arm/Group | Raltegravir 800 mg q.d. | Raltegravir 400 mg b.i.d.
Number analyzed (Participants) | 382 | 386
Participants | 318 | 343
Statistical Analysis 1: Comparison: Raltegravir 800 mg q.d. vs Raltegravir 400 mg b.i.d; Test type: Non-Inferiority or Equivalence — The 800 mg q.d. dosage was considered non-inferior to 400 mg b.i.d. if the lower bound of the 2-sided exact 95% CI for difference in response rate remained above -10%; p = 0.044, Miettinen and Nurminen; Mean Difference (Final Values) = -5.7, 95% CI 2-sided [-10.7 to -0.83]

2. Secondary Outcome: Number of Participants With HIV Ribonucleic Acid (RNA) <400 Copies/mL at 48 Weeks
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Raltegravir 800 mg q.d. | Raltegravir 400 mg b.i.d.
Number analyzed (Participants) | 382 | 386
Participants | 338 | 361
Statistical Analysis 1: Comparison: Raltegravir 800 mg q.d. vs Raltegravir 400 mg b.i.d; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.011, Miettinen and Nurminen; Mean Difference (Final Values) = -5.1, 95% CI 2-sided [-9.29 to -1.06]

3. Primary Outcome: Number of Participants With One or More Adverse Events at 48 Weeks
Time Frame: Week 48
Population: Data were analyzed for all randomized participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Raltegravir 800 mg q.d. | Raltegravir 400 mg b.i.d.
Number analyzed (Participants) | 382 | 388
Participants | 331 | 337
Statistical Analysis 1: Comparison: Raltegravir 800 mg q.d. vs Raltegravir 400 mg b.i.d; Test type: Superiority or Other; Miettinen and Nurminen; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-5.0 to 4.6]

4. Primary Outcome: Number of Participants Who Discontinued Due to an Adverse Event at 48 Weeks
Time Frame: Week 48
Population: Data were analyzed for all randomized participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Raltegravir 800 mg q.d. | Raltegravir 400 mg b.i.d.
Number analyzed (Participants) | 382 | 388
Participants | 4 | 3
Statistical Analysis 1: Comparison: Raltegravir 800 mg q.d. vs Raltegravir 400 mg b.i.d; Test type: Superiority or Other; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-1.3 to 2.0]

5. Secondary Outcome: Mean Change From Baseline to Week 48 in CD4 Cell Count
Time Frame: Baseline and Week 48
Population: Data were analyzed for all participants treated with study drug. Baseline values were carried forward for participants who discontinued treatment due to lack of efficacy.
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | Raltegravir 800 mg q.d. | Raltegravir 400 mg b.i.d.
Number analyzed (Participants) | 382 | 386
cells/mm^3 | 209.76 [194.6 to 224.9] | 196.20 [181.8 to 210.6]
Statistical Analysis 1: Comparison: Raltegravir 800 mg q.d. vs Raltegravir 400 mg b.i.d; Test type: Superiority or Other; t-test, 2 sided; Mean Difference (Net) = 13.56, 95% CI 2-sided [-7.29 to 34.40]

6. Secondary Outcome: Number of Participants With HIV RNA <50 Copies/mL at 96 Weeks
Description: As the study was terminated after the 48-week analysis, the planned secondary analyses for Week 96 were not performed.
Time Frame: Week 96
Population: The Week 96 data analysis was not performed.
Arm/Group | Raltegravir 800 mg q.d. | Raltegravir 400 mg b.i.d.
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Participants With HIV RNA <400 Copies/mL at 96 Weeks
Description: As the study was terminated after the 48-week analysis, the planned secondary analyses for Week 96 were not performed.
Time Frame: Week 96
Population: The Week 96 data analysis was not performed.
Arm/Group | Raltegravir 800 mg q.d. | Raltegravir 400 mg b.i.d.
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Mean Change From Baseline to Week 96 in CD4 Cell Count
Description: As the study was terminated after the 48-week analysis, the planned secondary analyses for Week 96 were not performed.
Time Frame: Baseline and Week 96
Population: The Week 96 data analysis was not performed.
Groups:
- Raltegravir 800 mg q.d.: Raltegravir 800 mg PO q.d. plus placebo to raltegravir PO b.i.d. plus one tablet of TRUVADA™ for 96 weeks
- Raltegravir 400 mg b.i.d.: Raltegravir 400 mg b.i.d. administered with TRUVADA™
Arm/Group | Raltegravir 800 mg q.d. | Raltegravir 400 mg b.i.d.
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Number of Participants With One or More Adverse Events at 96 Weeks
Description: As the study was terminated after the 48-week analysis, the planned secondary analyses for Week 96 were not performed.
Time Frame: Week 96
Arm/Group | Raltegravir 800 mg q.d. | Raltegravir 400 mg b.i.d.
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Number of Participants Who Discontinued Due to an Adverse Event at 96 Weeks
Description: As the study was terminated after the 48-week analysis, the planned secondary analyses for Week 96 were not performed.
Time Frame: Week 96
Arm/Group | Raltegravir 800 mg q.d. | Raltegravir 400 mg b.i.d.
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Overall Study
Arm/Group | Raltegravir 800 mg q.d. | Raltegravir 400 mg b.i.d.
Serious Adverse Events (participants affected / at risk) | 29/382 | 46/388
Other Adverse Events (participants affected / at risk) | 287/382 | 282/388
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raltegravir 800 mg q.d. (N=382) | Raltegravir 400 mg b.i.d. (N=388)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Retroperitoneal lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 4 (4)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Immune reconstitution syndrome (Immune system disorders) | 0 (0) | 1 (1)
Abscess intestinal (Infections and infestations) | 1 (1) | 0 (0)
Abscess jaw (Infections and infestations) | 1 (1) | 0 (0)
Anogenital warts (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 2 (2) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 1 (1)
Eye infection syphilitic (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2)
Histoplasmosis (Infections and infestations) | 0 (0) | 1 (1)
Meningitis aseptic (Infections and infestations) | 1 (1) | 0 (0)
Meningitis cryptococcal (Infections and infestations) | 1 (2) | 0 (0)
Meningitis viral (Infections and infestations) | 0 (0) | 1 (1)
Mycobacterium avium complex infection (Infections and infestations) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 1 (1) | 0 (0)
Perirectal abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0)
Post procedural pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Shigella infection (Infections and infestations) | 1 (1) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Multiple drug overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Penis injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anal cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Kaposi's sarcoma AIDS related (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Retroperitoneal neoplasm metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 2 (2) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 4 (4)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal colic (Renal and urinary disorders) | 2 (3) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Amenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Epididymitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raltegravir 800 mg q.d. (N=382) | Raltegravir 400 mg b.i.d. (N=388)
Lymphadenopathy (Blood and lymphatic system disorders) | 22 (23) | 21 (23)
Abdominal pain (Gastrointestinal disorders) | 13 (14) | 21 (27)
Diarrhoea (Gastrointestinal disorders) | 70 (81) | 70 (87)
Nausea (Gastrointestinal disorders) | 41 (47) | 54 (57)
Vomiting (Gastrointestinal disorders) | 24 (29) | 25 (36)
Fatigue (General disorders) | 25 (28) | 27 (30)
Pyrexia (General disorders) | 19 (23) | 26 (35)
Bronchitis (Infections and infestations) | 31 (32) | 28 (34)
Gastroenteritis (Infections and infestations) | 21 (23) | 14 (18)
Influenza (Infections and infestations) | 25 (28) | 36 (40)
Nasopharyngitis (Infections and infestations) | 40 (51) | 54 (70)
Sinusitis (Infections and infestations) | 16 (17) | 30 (36)
Upper respiratory tract infection (Infections and infestations) | 49 (64) | 54 (70)
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 (22) | 25 (32)
Back pain (Musculoskeletal and connective tissue disorders) | 23 (28) | 22 (25)
Dizziness (Nervous system disorders) | 36 (39) | 29 (35)
Headache (Nervous system disorders) | 58 (70) | 62 (87)
Depression (Psychiatric disorders) | 22 (22) | 23 (25)
Insomnia (Psychiatric disorders) | 18 (18) | 22 (22)
Cough (Respiratory, thoracic and mediastinal disorders) | 38 (40) | 30 (41)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 15 (19) | 20 (23)
Rash (Skin and subcutaneous tissue disorders) | 23 (26) | 23 (27)
Hypertension (Vascular disorders) | 11 (11) | 22 (22)

LIMITATIONS AND CAVEATS:
The study was terminated before the 96-week efficacy analysis. Adverse event data were collected for the entire treatment period up to a maximum of Week 108, which defines the Overall Study period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Twenty-four months after completion of this study or after publication of the multicenter results, an investigator may publish the results for their study site independently. The sponsor must have the opportunity to review all proposed publications or presentations regarding the study 60 days before submission.